CLINICAL TRIAL: NCT04129255
Title: IMMUNeOCT Study: Octreotide LAR in the Induction of Immunologic Response in Patient With Neuroendocrine Tumors: an Interventional Pharmacological Study
Brief Title: Octreotide LAR in the Induction of Immunologic Response in NENs Patients
Acronym: CSMS99
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Salvatore Tafuto, MEDICAL DOCTOR, National Cancer Institute, Naples
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNeOCT
Record Dates: First submitted 2019-08-27; First posted 2019-10-16 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Tumors
Keywords: Octreotide; neuroendocrine tumors; immunological response
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Octreotide; Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OCTREOTIDE LONG-ACTING RELEASE (OCT LAR) (Other): OCT LAR is already registered By FDA for USA, by EMA for Europe and , also, by AIFA for Italy.
  Interventions: Drug: Octreotide Acetate

INTERVENTIONS:
Drug: Octreotide Acetate — administration every 28 days
  Other Names: Somatostatin analog

SUMMARY:
Evaluating the impact of OCTREOTIDE LAR on the immune response by studying Regulatory T-cell (T-Reg) and Myeloid-derived suppressor cells (MDSC) and the immunoregulatory cell population in peripheral blood of NET G1 / G2 patients treated with Octreotide LAR

DETAILED DESCRIPTION:
MDSCs and T-Regs will be evaluated at baseline pre-treatment with octreotide, after 15 days, at three and at six months and before each octreotide LAR administration for 12 months. MDSC cells will be detected by surface receptors LIN-, CD11b, CD14, CD15, CD33, CD124-IL4-Ra, CD184-CXCR4, CD279-PD1, HLA-DR and T-reg cells from CD3, CD4, CD8 receptors , CD25, CD39, CD45RA, CD45R0, CD62L, CD127, CD152-CTLA-4, CD184-CXCR4, CD278-ICOS, CD279-PD-1. Briefly, CD4 + cells will be separated by negative selection, using the mixture of human CD4 antibodies. Octreotide is currently a registered drug to the FDA, EMA and AIFA with the indication for the treatment of well and moderately differentiated NETs functioning and not working on the front line. .

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures or treatment, as confirmation of the patients awareness and willingness to comply with the study requirements.
* Patients ≥18 years of age.
* Patients with histologically confirmed well and moderately differentiated Neuroendocrine Tumors with Ki67 ≤ 20% (Ki67 must be quantified in percentage) and candidates for treatment with octreotide.
* ECOG performance status (PS) of 0-2.
* At least 28 days since prior the last radiation therapy or surgery.
* Estimated life expectancy of ≥12 weeks.

Exclusion Criteria:

* Patients < 18 years of age.
* According to the current SmPC of the prescribed drug agent.
* Previuos treatment with octreotide.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would prevent the patient from meeting the study requirements.
* Serious active infection requiring i.v. antibiotics and/or hospitalization at study entry.
* Patients who are treated with any medicinal product that contraindicates the use of the study drug, may interfere with the planned treatment, affects patient compliance or puts the patient at high risk for treatment-related complications.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start. Women of childbearing potential (defined as inferior to 2 years after last menstruation and not surgically sterile) not using effective, non hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patients with meningeal carcinomatosis
* Patients with known positive HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Exploring the changes in immune-regulatory cells induced by OCT LAR | 6 months
  The primary objective of the project is to evaluate changes in immune-regulatory cells induced by OCT LAR from baseline to month 6. Therefore, we will observe the impact of OCTREOTIDE LAR on the immune response by studying T-Reg and MDSC and the immunoregulatory cell population in peripheral blood of patients with neuroendocrine tumors G1 / G2 treated with OCT LAR.

SECONDARY OUTCOMES:
Outcome | 3 months (PFS - ORR)
  Objective response rate according to RECIST.
  Progression-free survival (PFS), defined as the time (days) from start date of octreotide to date of first documented disease progression or death due to any cause, if death occurs before progression is documented.
  Progression-free survival as the time (days) from start date of OCT to date of first PD or death due to any cause; Safety :number of patients presenting AE during treatment and observation period (CTCAE v.4)
safety assessment | 1 month (safety)
  Safety profile according to CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Tafuto, MD, Principal Investigator — NCI Naples
Locations (1):
- Istitute Nazionale Tumori - Fondazione G. Pascale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No